CLINICAL TRIAL: NCT04750447
Title: Safety and Efficacy of an Ab Interno Gelatin Stent (XEN63) With or Without Mitomycin C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prism Eye Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Iqbal Ahmed, Principal Investigator, Prism Eye Institute
Other Study IDs: 1035
Record Dates: First submitted 2021-02-09; First posted 2021-02-11 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Open Angle Glaucoma: Patients aged 30-90 Primary open angle glaucoma on maximum tolerated medical therapy Going to receive XEN63 ab interno gelatin stent with or without MMC in study eye ± cataract surgery
  Interventions: Device: XEN 63

INTERVENTIONS:
Device: XEN 63 — The Xen gelatin microstent (Allergan, CA, USA) is a 6mm gelatin tube used in microinvasive glaucoma surgery (MIGS) to create a bleb. A bleb is a fluid filled blister located in the tissue covering the white portion of the eye (the conjunctiva) created after glaucoma surgery. The bleb allows the eye pressure (intraocular pressure - IOP) to be lowered by bypassing the natural pathways by which the fluid called aqueous leaves the eye and redirecting it towards the bleb to be absorbed by other pathways. Amongst the main advantages of this device is the ability to create a bleb without disrupting tissue unlike other methods of glaucoma surgery (e.g., trabeculectomy). This decreases the amount of wound healing and scarring, and potentially limiting bleb failure.

SUMMARY:
The Xen gelatin microstent (Allergan, CA, USA) is a 6mm hydrophobic, bleb-forming microinvasive glaucoma surgery (MIGS).1 Creation of a filtering bleb through the gel stent and under the conjunctiva lowers intraocular pressure (IOP) by bypassing the natural outflow pathway of aqueous. Currently three Xen models have been developed: 45, 63, and 140 um internal lumen diameters.2 XEN45 ab interno gelatin stent was the first to be approved for clinical use in Canada.3 A recent retrospective cohort study showed comparable safety and risk of failure to trabeculectomy.4 Amongst the main advantages of this device is the ability to create a bleb without dissecting and disrupting tissue, thus decreasing the amount of wound healing and potentially limiting bleb failure. Recently, the XEN63 ab interno gelatin stent was approved by Health Canada for clinical use in Canada. Being a new device, to date, no study has examined the effect of XEN63 ab interno gelatin stent on anti-glaucoma drops burden and IOP. The aim of this study is to investigate the safety and efficacy of the XEN63 ab interno gelatin stent to provide insights for ophthalmologists who will want to add this technique to their practice.

DETAILED DESCRIPTION:
• This is a prospective, single-arm, open-label clinical trial designed to demonstrate the safety and IOP-lowering effectiveness of XEN 63. Approximately 29 patients who are scheduled to undergo glaucoma surgery with XEN63 implantation will be enrolled and followed for up to 12 months postoperatively. Enrollees will follow the standard of care visits (pre-op, post-op day 1, post-op week 1 and post op month 1) where they will undergo a full eye exam (visual acuity, refraction, slit lamp exam and intraocular pressure measurement). In addition to the standard of care visit, enrollees will have 2 additional visits (post-op month 6 and post-op month 12) where they will undergo a full eye exam. Additional tests include a Visual Field assessment and Endothelial cell count on their pre-op visit, post-operative month visit 6 and post-op month 12 visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-90 Primary open angle glaucoma on maximum tolerated medical therapy Going to receive XEN63 ab interno gelatin stent with or without MMC in study eye ± cataract surgery

Exclusion Criteria:

* Other forms of glaucoma
* Previous glaucoma shunt/valve in the target quadrant of study eye
* Presence of conjunctival scarring, prior conjunctival surgery or other conjunctival pathologies (e.g., pterygium) in the target quadrant of study eye
* Active inflammation (e.g., blepharitis, conjunctivitis, keratitis, uveitis), active iris neovascularization or neovascularization of the iris within six months of the surgical date
* Presence of anterior chamber intraocular lens, intraocular silicone oil, vitreous present in the anterior chamber, impaired episcleral venous drainage (e.g., Sturge-Weber or nanophthalmos or other evidence of elevated venous pressure)
* Known or suspected allergy or sensitivity to drugs required for the surgical procedure or any of the device components (e.g., porcine products or glutaraldehyde), history of dermatologic keloid formation.
* Prior CPC, corneal graft (PKP, DALK, DSAEK, DMEK)
* Other forms of combined surgery (cornea, retina) besides cataract surgery

Ages: 30 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo Xen 63 implantation for open angle glaucoma with or without cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2023-06-09 (Estimated); Study Completion 2023-06-09 (Estimated)

PRIMARY OUTCOMES:
Complete Success | 1 month post op to post op month 12
  Intraocular Pressure: 6-17 mmHg and on no glaucoma medications at least 1 month after surgery with no reoperation using the Goldmann Applanation Tonometer..
Absence of complications | post op day 1 to post op month 12
  Absence of the following complications as reported during slitlamp examination:
  i. Starting after POM1: shallow AC w/ iridocorneal touch, any hyphema, corneal edema, choroidal effusion, malignant glaucoma, dellen/non-healing epithelial defect, ptosis, diplopia.
  ii. At any point: additional glaucoma surgery, loss of light perception vision, vitreous hemorrhage, ≥2mm hyphema, hypotony maculopathy, implant migration/blockage/exposure/extrusion, macular edema, choroidal effusion/hemorrhage requiring drainage, suprachoroidal hemorrhage, retinal detachment, blebitis/endophthalmitis
Qualified Success | post op month 1 to post op month 12
  a. 'Complete success' criteria except that Intraocular Pressure (IOP) can be above IOP thresholds, and then reduced to within the 'Complete criteria' by medications or laser in 3 visits or less as measured by Goldmann Applanation Tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Ahmed, MD, Principal Investigator — Prism Eye Institute
Locations (1):
- Prism Eye Institute, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conlon R, Saheb H, Ahmed II. Glaucoma treatment trends: a review. Can J Ophthalmol. 2017 Feb;52(1):114-124. doi: 10.1016/j.jcjo.2016.07.013. Epub 2016 Nov 17. PMID 28237137
- [Background] Green W, Lind JT, Sheybani A. Review of the Xen Gel Stent and InnFocus MicroShunt. Curr Opin Ophthalmol. 2018 Mar;29(2):162-170. doi: 10.1097/ICU.0000000000000462. PMID 29319544
- [Background] Schlenker MB, Gulamhusein H, Conrad-Hengerer I, Somers A, Lenzhofer M, Stalmans I, Reitsamer H, Hengerer FH, Ahmed IIK. Efficacy, Safety, and Risk Factors for Failure of Standalone Ab Interno Gelatin Microstent Implantation versus Standalone Trabeculectomy. Ophthalmology. 2017 Nov;124(11):1579-1588. doi: 10.1016/j.ophtha.2017.05.004. Epub 2017 Jun 7. PMID 28601250